CLINICAL TRIAL: NCT01949272
Title: Optimization of PEEP for Alveolar Recruitment in ARDS
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Collaborators: Melun Hospital Intensive Care Unit (Unknown)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, MD, Hopital of Melun
Other Study IDs: OPERA
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: ARDS
Keywords: ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ARDS: ARDS patients achieving stades II and III of Berlin 2011 Classification
  Interventions: Device: esophageal pressure mesurement

INTERVENTIONS:
Device: esophageal pressure mesurement — "EXPRESS study" ventilatory setting the optimization of PEEP with esophageal pressure mesurement

SUMMARY:
Actual setting of PEEP in ARDS is based on tables linked to FiO2, or respiratory system plateau pressure (e.g EXPRESS Study) or set regarding esophageal pressure mesurement and transpulmonary pressure calculation. Opera study should confirm if a setting approach based on esophageal pressure is helpfull for any ARDS patient in ICU without deleterious side-effect.

ELIGIBILITY:
Inclusion Criteria:

* ARDS Stades 2 and 3 with invasive ventilation (EXPRESS settings) within 3 to 12 hours

Exclusion Criteria:

* less 18 years, pregnancy, intracardiac shunt, esophageal catheter cons-indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients achievinf definition of ARDS stades II and III of Berlin Classification
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | 24 hours

SECONDARY OUTCOMES:
Vd/Vt ratio | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Monchi, MD, Study Director — Melun Hospital ICU
Locations (1):
- Melun Hospital ICU, Melun, France